CLINICAL TRIAL: NCT04308564
Title: Constitution d'Une Collection d'Echantillons Biologiques Associee a Une Base de Donnees de Patients Possedant Des Anticorps Antiphospholipides
Brief Title: Laboratory and Clinical Data in Antiphospholipid Patients
Acronym: APSregistry
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Pr Denis WAHL, Head of Vascular Medicine Division, Principal Investigator, Professor of Vascular Medicine, Central Hospital, Nancy, France
Other Study IDs: 2019-A02058-49
Record Dates: First submitted 2020-03-09; First posted 2020-03-16 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Antiphospholipid Syndrome
Keywords: antiphospholipid antibodies
MeSH Terms: conditions — Antiphospholipid Syndrome | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — DNA, plasma and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood test — Blood test for the identification of biomarkers

SUMMARY:
To constitute a registry of antiphospholipid antibodies positive-patients

DETAILED DESCRIPTION:
An international web-based application, the REDCap (Research Electronic Data Capture), captures data on patient demographics, aPL-related clinical and laboratory characteristics, and medications. The inclusion criteria are: a) age between 18 and 60 years; and b) persistent (at least 12 weeks apart) aPL-positivity within 12 months prior to screening; positivity is defined as anticardiolipin antibodies (aCL) IgG/M/A (> 40 GPL/MPL/APL, medium-to-high titer, and/or greater than the 99th percentile), anti-β2-glycoprotein-I (aβ2GPI) IgG/M/A (> 40 units, medium-to-high titer), positive lupus anticoagulant (LA) test based on International Society on Thrombosis and Hemostasis and other current guidelines. Patients are followed every 12 ± 3 months with clinical data and blood collection. Blood drawn is done at inclusion and every year.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 60 years;
* persistent (at least 12 weeks apart) aPL-positivity within 12 months prior to screening

Exclusion Criteria:

* no inform consent
* impossible follow up
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Antiphospholipid antibodies positive-patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2030-04-01 (Estimated); Study Completion 2031-04-01 (Estimated)

PRIMARY OUTCOMES:
Thrombosis | Up to 10 years
  Rate of thrombosis

SECONDARY OUTCOMES:
Bleeding | Up to 10 years
  Rate of bleeding

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHRU de Lille, Lille
  - CHRU de Nancy, Nancy

IPD SHARING:
Plan to Share IPD: Undecided